CLINICAL TRIAL: NCT04281888
Title: Mortality Associated Parameters With Inflammatory Anemia in Patients With Sepsis Admitted to the Intensive Care Unit and Blood Transfusion Effect
Brief Title: Inflammatory Anemia Associated Parameters in Septic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Mohamed Ahmed, Hematologist, Assiut University
Other Study IDs: Heba
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Inflammatory Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
1. To observe the changes in the inflammatory anemiaassociated parameters of patients with sepsis in the early stage of intensive care unit (ICU) admission.
2. To evaluate their association with 28-days mortality
3. To evaluate the effect of blood transfusion on these parameters and the survival of the studied patients

DETAILED DESCRIPTION:
Anemia is one of the most common complications in patients with sepsis in the intensive care unit (ICU), as well as sepsis is a major cause of high mortality in ICU. Studies demonstrated that sepsis-related anemia can be caused by fluid loading related hemodilution, iatrogenic blood loss, decreases in iron supply, erythropoietin (EPO) production and erythrocyte lifespan .

However, sepsis related anemia has been demonstrated to be associated mainly with inflammation (i.e., "anemia of inflammation"). Anemia of inflammation is usually a mild to moderately severe anemia (hemoglobin rarely < 8 g/dL) . It develops in the setting of infection, inflammatory disease or malignancy, together with low serum iron despite adequate systemic iron stores, decreased serum transferrin, normal size of erythrocytes and hemoglobin content or mildly decreased size and hemoglobin content of erythrocytes if the inflammatory disease is longstanding .

Impaired iron homeostasis and the suppressive effects of proinflammatory cytokines on erythropoiesis, together with alterations in the erythrocyte membrane that impair its survival may result, ultimately, in inflammation-associated anemia .

Hepcidin is a key regulator of inflammation-associated anemia. Hepcidin reduces the iron level in plasma through:

1. direct inhibition of intestinal absorption of iron.
2. promotion of iron storage in macrophages by down regulating expression of ferroprotein in intestinal mucosae and macrophages.

Increased interleukin-6 (IL-6) in patients with sepsis can induce an abruptly increased synthesis of hepcidin, causing decreased plasma iron. Plasma iron can be depressed by inflammation markedly (more than 50%) and rapidly ( with in 24 hrs). Also, the interaction between inflammation and iron metabolism may interfere with other inflammatory anemia associated parameters and complicate iron metabolism in patients with sepsis.

Typically, plasma ferritin (which stores iron) is reduced in iron deficiency anemia but can increase in the acute phase of sepsis. Anemia usually results in an increased synthesis of EPO in kidneys in minutes to hours, but the response to EPO is blunted in patients with sepsis . The soluble transferrin receptor (sTfR), an early and sensitive biomarker for diagnosing iron deficiency , is particularly useful for identification of concomitant iron deficiency in patients with inflammation. The sTfR is not affected by inflammation, which is a significant advantage over other biomarkers. Plasma sTfR reflects the degree of iron availability for cells, whereas plasma ferritin reflects iron storage. Hence, the ratio of sTfR to log ferritin (hereafter termed "sTfR/log ferritin") provides the efficacy of sTfR alone or ferritin alone in the diagnosis of iron deficiency. These cytokines have the propensity to promote iron restricted erythropoiesis, characterized by functional rather than absolute iron deficiency, occurring secondary to dysregulation of iron metabolism.

Associations among inflammatory cytokines, EPO, and anemia in critically ill septic patients remain unclear.

The inflammatory anemia-associated parameters mentioned above may change with the severity of inflammation in patients with sepsis. The sensitivity and specificity of these parameters can be modified if inflammation and iron deficiency are present concomitantly. This may complicate the diagnosis, evaluation, and treatment of inflammatory anemia.

Hence, a better understanding of changes in the inflammatory anemia and associated parameters in patients with sepsis at the early stage of ICU admission is needed urgently. In addition, although severe anemia is associated with adverse outcomes in critical illness, a lowered plasma iron is part of the natural defense against pathogens.

EPO has also been demonstrated to exert protective effects in the kidneys and lungs of mice with sepsis, but EPO deficiency contributes to anemia development in patients with sepsis. As a result of these effects, inflammatory anemia-associated parameters have been speculated to be associated with the prognosis of patients with sepsis , but relevant studies are lacking

ELIGIBILITY:
Inclusion Criteria:

1-patients meeting diagnostic criteria of sepsis and hemoglobin level less than 10 g/dl 2-patients admitted to the intensive care unit Exclusion Criteria

1. patients less than18 years of age.
2. patients have chronic liver dysfunctions or chronic kidney disease resulting from different causes.
3. patients with known iron related diseases (e.g., hemochromatosis), immunologic diseases or malignancies upon hospital admission; all types of anemia (aplastic, iron deficiency, hemolytic, megaloblastic).
4. patients with overt blood loss (e.g., gastrointestinal bleeding) upon admission and during the ICU stay.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients in ICU with sepsis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-03-20 (Estimated); Primary Completion 2021-03-20 (Estimated); Study Completion 2021-05-20 (Estimated)

PRIMARY OUTCOMES:
The relation between level of hepcidin, interleukin-6 and hemoglobin with 28-days mortality in 100 ICU septic patients | Baseline
  Hepicidin level will be measured in day 1,3 and 7 of ICU admission as well as interleukin-6 and hemoglobin and the relation between their level and survival of the studied patients will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Yousreiya A Ahmad, Professor, Study Director — Assuit University Hospital

REFERENCES:
- [Background] Ganz T, Nemeth E. Iron homeostasis in host defence and inflammation. Nat Rev Immunol. 2015 Aug;15(8):500-10. doi: 10.1038/nri3863. Epub 2015 Jul 10. PMID 26160612
- [Background] Hegde A. Approach to an Anemic Critically Ill Patient. Indian J Crit Care Med. 2019 Sep;23(Suppl 3):S178-S180. doi: 10.5005/jp-journals-10071-23247. PMID 31656373
- [Background] Weiss G, Ganz T, Goodnough LT. Anemia of inflammation. Blood. 2019 Jan 3;133(1):40-50. doi: 10.1182/blood-2018-06-856500. Epub 2018 Nov 6. PMID 30401705